CLINICAL TRIAL: NCT04513275
Title: Research on Accurate Prediction of Long-term Medication Use for Schizophrenia Based on Cognitive Function
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: PLFSBC
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Non-medicine Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- schizophrenia patient group: Schizophrenia patients with first episode and disease duration of 5, 10, 20, and 30 years
  Interventions: Drug: non-medicine intervention

INTERVENTIONS:
Drug: non-medicine intervention — rating by MCCB only one time
  Other Names: rating by MATRICS Consensus Cognitive Battery,MCCB

SUMMARY:
Chinese version of the cognitive function test of schizophrenia (MCCB) . To explore a predictive model for long-term medication use in patients based on cognitive function

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia patients with first episode and disease duration of 5, 10, 20, and 30 years _Meet the diagnostic criteria for schizophrenia in ICD-10

Exclusion Criteria:

* Other people with mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Schizophrenia patients with first episode and disease duration of 5, 10, 20, and 30 years
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Score of MATRICS Consensus Cognitive Battery | 1 day (only one time)

IPD SHARING:
Plan to Share IPD: No